CLINICAL TRIAL: NCT05222009
Title: Adding G-CSF in Patients With Anti-PD-1-axis Therapy-resistant Recurrent or Metastatic
Brief Title: G-CSF in Patients With Anti-PD-1-axis Therapy-resistant Recurrent or Metastatic Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ming-Yuan Chen, Chief physician, Proffessor, Sun Yat-sen University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC-CMY-2021-1214
Record Dates: First submitted 2022-01-24; First posted 2022-02-03 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: Granulocyte Colony-Stimulating Factor; PD-1 Inhibitor
MeSH Terms: interventions — pegylated granulocyte colony-stimulating factor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- G-CSF arm1 (Experimental): PD-1 inhibitor resistance regimen+ G-CSF 3mg
  Interventions: Drug: PEG-rhG-CSF
- G-CSF arm2 (Experimental): PD-1 inhibitor resistance regimen+ G-CSF 6mg
  Interventions: Drug: PEG-rhG-CSF

INTERVENTIONS:
Drug: PEG-rhG-CSF — PEG-rhG-CSF, 3mg, D1, Q3W, subcutaneous injection, until stop using PD-(L)1 inhibitor, progressive disease (PD) or unacceptable toxicity. Meanwhile, the original maintenance regimen--PD-(L)1 inhibitor ± VEGFR/EGFR TKI/Ab--continues.
  Arms: G-CSF arm1
Drug: PEG-rhG-CSF — PEG-rhG-CSF, 6mg, D1, Q3W, subcutaneous injection, until stop using PD-(L)1 inhibitor, progressive disease (PD) or unacceptable toxicity. Meanwhile, the original maintenance regimen--PD-(L)1 inhibitor ± VEGFR/EGFR TKI/Ab--continues.
  Arms: G-CSF arm2

SUMMARY:
Recurrence and metastasis are the main causes of treatment failure of NPC. Immunotherapy is an emerging cancer treatment method, which has less adverse reactions and longer duration compared with chemotherapy. At present, there are a large number of PATIENTS with anti-PD-1 resistance in clinical practice, who are faced with a significant decline in the efficacy of anti-PD-1 after treatment. However, without the synergistic effect of anti-PD-1, survival after chemotherapy alone will be significantly shortened. how to improve the efficacy of immunotherapy rechallenge so that a large number of potential patients can benefit from immunotherapy is an urgent problem to be solved at present.

Studies have shown that G-CSF can significantly increase the proportion of effector cells dominated by CD4+ T cells, improve the diversity of peripheral blood TCR, thus regulate the immune status of tumor patients. Therefore, G-CSF may have a synergistic effect on anti-PD-1. This study intends to explore whether the addition of G-CSF can restore the efficacy of anti-PD-1 in drug-resistant NPC patients through a prospective clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female; 18-75 years of age.
2. Subjects diagnosed with pathological confirmed non-keratinizing (WHO-II/III) metastatic NPC, or subjects with recurrent NPC that is unfit for local treatment
3. Received prior treatment with platinum agents and PD-(L)1 inhibitors.
4. Developed acquired resistant (AR) to PD-(L)1 inhibitors following the anti-PD-1/L1 or combined with anti-target agent (VEGFR/EGFR TKI/Ab) maintenance therapy. (AR defined as disease progression after partial or complete response).
5. Patients must have at least 1 lesion that is measurable using RECIST v1.1 criteria.
6. ECOG performance status of 0 or 1.
7. Have recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to any anti-tumor therapy 4 weeks earlier. Except for hair loss, hair color change, nail change, fatigue, etc., which do not pose safety risks to subjects.
8. Life expectancy more than 12 weeks.
9. Patients must have adequate organ function (without blood transfusion, without growth factor or blood components support within 14 days before enrollment) as determined by:

   Absolute neutrophil count (ANC) ≥1.5×109/L; Platelet count ≥ 75×109/L; Hemoglobin ≥ 9 g/dL; serum total bilirubin (TBIL) ≤1.5 times the upper limit of normal (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×upper limit of normal (ULN), (for subjects with liver metastases, TBIL ≤3×ULN ; ALT and AST≤5×ULN); Creatinine ≤1.5×ULN or creatinine clearance rate≥50 ml/min (Cockcroft-Gault formula); serum albumin ≥28 g/L; INR, APTT≤1.5 x ULN.
10. Female subjects agree not to be pregnant or lactating from beginning of the study screening through at least 3 months after receiving the last dose of study treatment. Both men and women of reproductive potential must be willing and able to employ a highly effective method of birth control/contraception to prevent pregnancy.
11. Be willing and able to provide written informed consent/assent for the trial.

Exclusion Criteria:

1. Known history of any ≥ grade 3 immune-related toxicity.
2. Known history of hypersensitivity to any components of the PEG-rhG -CSF formulation.
3. Received G-CSF concurrent with anti-PD-(L)1 antibody combined with anti-target agent (VEGFR/EGFR TKI/Ab) maintenance therapy. (Patients who received G-CSF to prevent and treat febrile neutropenia secondary to chemotherapy are permitted)
4. Prior chemotherapy, targeted small molecule therapy, or radical therapy within 2 weeks prior to Study Day 1
5. Diagnosed and/or treated additional malignancy within 5 years of enrollment, with the exception of curatively-treated basal cell or squamous cell carcinoma of the skin, and/or curatively-resected in situ cervical and/or breast carcinoma.
6. Concurrent medical condition requiring the use of immunosuppressive medications, or immunosuppressive doses of systemic or absorbable topical corticosteroids. Doses > 10 mg/day prednisone or equivalent are prohibited within 2 weeks before study drug administration.
7. Active central nervous system metastases and/or carcinomatous meningitis
8. Severe, uncontrolled angiocardiopathy (heart failure > class II NYHA, unstable angina, myocardial infarction within past 1 year, supraventricular or ventricular arrhythmia which need medical intervention, or QT interval male ≥ 450 ms, female ≥ 470 ms.).
9. History of non-infectious pneumonitis that required steroids or current pneumonitis
10. Active infection requiring systemic therapy
11. Be known to have active tuberculosis.
12. Human immunodeficiency virus (HIV) positive
13. Hepatitis B or C positive
14. Live vaccine within 30 days of planned start of study drug
15. Underlying medical condition that, in the Investigator's opinion, would increase the risks of study drug administration or obscure the interpretation of toxicity determination or adverse events.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-01-24 (Estimated); Primary Completion 2022-11-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
ORR | 1 year
  Defined as the proportion of patients whose tumors shrink to complete response (CR) or partial response (PR) and remain for a certain period of time according to RECIST 1.1

SECONDARY OUTCOMES:
The proportion of patients who achieved disease control | 1 year
  Defined as the proportion of subjects who achieve CR+PR+stable disease (SD) for at least 4 weeks according to RECIST 1.1.
The proportion of patients who achieved clinical benefit | 1 year
  Defined as maintaining the efficacy of CR+PR+SD for at least 6 months according to RECIST 1.1.
Duration of response | 1 year
  Defined as the time from the first assessment of CR and PR to the first assessment of PD or death caused by any cause according to RECIST 1.1.
median progression-free survival | 1 year
  Defined as the period from the start of enrollment until disease progression or death from any cause.
Adverse events | 1 year
  assessed by NCI-CTC5.0 standard

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nasopharyngeal Carcinoma, Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China